CLINICAL TRIAL: NCT02973386
Title: Randomized Trial of Concurrent Cisplatin Chemoradiotherapy Plus Capecitabine Adjuvant Chemotherapy vs Concurrent Cisplatin Chemoradiotherapy Alone for Patients With Local Advanced Nasopharyngeal Carcinoma at High Risk of Distant Metastasis
Brief Title: Prognostic Analysis of Concurrent Chemoradiotherapy With/Without Adjuvant Chemotherapy for Locally Advanced NPC Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCRT-AC-HRDM-NPC
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Local Advanced High Risk Nasopharyngeal Carcinoma
Keywords: Local advanced; High Risk; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent chemoradiation + adjuvant chemotherapy (Experimental): IMRT combine with cisplatin concurrent chemotherapy plus capecitabine adjuvant chemotherapy
  Interventions: Drug: IMRT combine with cisplatin concurrent chemotherapy plus capecitabine adjuvant chemotherapy
- Concurrent chemoradiation (Active Comparator): IMRT combine with cisplatin concurrent chemotherapy
  Interventions: Drug: IMRT combine with cisplatin concurrent chemotherapy

INTERVENTIONS:
Drug: IMRT combine with cisplatin concurrent chemotherapy — Patients in the control arm received radical radiotherapy with IMRT, and cisplatin (100mg/m2 on day 1 and day 22) during RT.
  Arms: Concurrent chemoradiation
Drug: IMRT combine with cisplatin concurrent chemotherapy plus capecitabine adjuvant chemotherapy — Patients in the experimental arm received radical radiotherapy with IMRT, and cisplatin (100mg/m2 on day 1 and day 22) during RT,followed by adjuvant chemotherapy with oral capecitabine(1000mg/m2/ twice a day for 14 days)every three weeks for eight cycles at 4 weeks later after RT.
  Arms: Concurrent chemoradiation + adjuvant chemotherapy

SUMMARY:
This is a randomized,controlled,prospective phase III clinical trial. The purpose of this study is to evaluate acute toxicity and efficacy of concurrent cisplatin chemoradiation with or without capecitabine as adjuvant chemotherapy in Local Advanced Nasopharyngeal Carcinoma at High Risk of Distant Metastasis.Exploring an Individualized comprehensive treatment plan which is reasonable,effective,low toxicity and fitting with Modern radiotherapy techniques for Local Advanced Nasopharyngeal Carcinoma at High Risk of Distant Metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma(WHO II/III)
* Clinical stage III~IVb(UICC/AJCC 7th)
* No distant metastasis
* Karnofsky Performance Status Scale≥70
* WBC count ≥ 4×109/L, neutrophil differential count≥ 1.5×109/L, Hemoglobin ≥ 90g/L, platelet count ≥ 100×109/L
* ALT or AST ≤2.5×ULN,bilirubin ≤2.5×ULN, Serum creatinine ≤1.5×ULN or Serum creatinine clearance≥60ml/min
* Sign the informed consent.

Exclusion Criteria:

* Angle of sexual squamous cell carcinomas and basal cell layout, squamous cell carcinomas
* Younger than 18 years old or older than 70 years old
* Are receiving other drugs treanment
* kidney disease
* Have suffered from other tumor or now suffering from other tumor
* Have recieved chemotherapy or radiotherapy
* Pregnancy or lactation
* unstable heart disease need timely treatment
* Severe cerebrovascular disease/canker/psychosis/uncontrolled diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2025-12 (Actual)

PRIMARY OUTCOMES:
Distant metastasis-free survival | Five year
  Defined as the time from date of recruitment to documented distant metastasis or death from any cause.

SECONDARY OUTCOMES:
Failure-free survival | Five year
  Defined as the time from date of recruitment to documented relapse or death from any cause.
Locoregional relapse-free survival | Five year
  Defined as the time from date of recruitment to documented locoregional relapse or death from any cause.
Overall survival | Five year
  Defined as the time from date of recruitment to death from any cause.
Acute toxicity | three months after corresponding treatment
  Acute toxicities were graded using the Common Toxicity Criteria for Adverse Events version 4.0 (CTCAE v4.0) for chemotherapy-specific toxicities, and the Radiation Therapy Oncology Group (RTOG) radiation morbidity scoring criteria for radiotherapy-specific toxicities.
Late toxicity | Five year
  Late toxicities were assessed annually using the RTOG radiation morbidity scoring criteria.

CONTACTS AND LOCATIONS:
Overall Officials: zhao chong, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn